CLINICAL TRIAL: NCT03394482
Title: Interventional, Randomized, Open-label, Three-group, Two-sequence Crossover, Single-dose, Bioequivalence Study of Lu AF35700 in Healthy Subjects Comparing the 5, 10 and 20 mg Commercial Tablet (Test) to the 5, 10 and 20 mg Clinical Tablet (Reference)
Brief Title: Bioequivalence Study of Lu AF35700
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 17481A; 2017-001335-39 (EudraCT Number)
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Healthy
MeSH Terms: interventions — Lu AF35700

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Lu AF35700 5 mg clinical formulation (Experimental)
  Interventions: Drug: Lu AF35700 5 mg clinical formulation
- Lu AF35700 5 mg commercial formulation (Experimental)
  Interventions: Drug: Lu AF35700 5 mg commercial formulation
- Lu AF35700 10 mg clinical formulation (Experimental)
  Interventions: Drug: Lu AF35700 10 mg clinical formulation
- Lu AF35700 10 mg commercial formulation (Experimental)
  Interventions: Drug: Lu AF35700 10 mg commercial formulation
- Lu AF35700 20 mg clinical formulation (Experimental)
  Interventions: Drug: Lu AF35700 20 mg clinical formulation
- Lu AF35700 20 mg commercial formulation (Experimental)
  Interventions: Drug: Lu AF35700 20 mg commercial formulation

INTERVENTIONS:
Drug: Lu AF35700 5 mg clinical formulation — Lu AF35700 tablets 5 mg oral single dose
  Arms: Lu AF35700 5 mg clinical formulation
Drug: Lu AF35700 5 mg commercial formulation — Lu AF35700 tablets 5 mg oral single dose
  Arms: Lu AF35700 5 mg commercial formulation
Drug: Lu AF35700 10 mg clinical formulation — Lu AF35700 tablets 10 mg oral single dose
  Arms: Lu AF35700 10 mg clinical formulation
Drug: Lu AF35700 10 mg commercial formulation — Lu AF35700 tablets 10 mg oral single dose
  Arms: Lu AF35700 10 mg commercial formulation
Drug: Lu AF35700 20 mg clinical formulation — Lu AF35700 tablets 20 mg oral single dose
  Arms: Lu AF35700 20 mg clinical formulation
Drug: Lu AF35700 20 mg commercial formulation — Lu AF35700 tablets 20 mg oral single dose
  Arms: Lu AF35700 20 mg commercial formulation

SUMMARY:
The purpose of this study is to establish bioequivalence of Lu AF35700 between the clinical formulation and the commercial formulation for three tablet strengths; 5, 10 and 20 mg

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged ≥18 and ≤55 years
* Body Mass Index (BMI) of ≥18.5 and ≤32 kg/m2
* Subject must be in good general health as assessed using medical history, clinical laboratory tests, and physical examination

Exclusion Criteria:

* The subject must not be of childbearing potential (if a woman) or should use contraception, be surgically sterilized or not be sexually active (both sexes). Women must not be pregnant or lactating
* The subject must not be a CYP2D6 or a CYP2C19 poor metaboliser
* The subject has previously been dosed with Lu AF35700

Other protocol defined inclusion and exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
AUC0-72h of Lu AF35700 | zero to 72 hours
  Area under the Lu AF35700 plasma concentration-time curve from zero to 72 hours post-dose (AUC0-72h)
Cmax of Lu AF35700 | zero to 72 hours
  Maximum observed plasma concentration (Cmax) of Lu AF35700

SECONDARY OUTCOMES:
Tmax of Lu AF35700 | zero to 72 hours
  Time to occurance of Cmax of Lu AF35700
AUC0-t of Lu AF35700 | zero to time of the last quantifiable plasma concentration
  Area under the Lu AF35700 concentration-time curve from zero to time of the last quantifiable plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H.Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- Covance, Leeds, United Kingdom